CLINICAL TRIAL: NCT05904912
Title: Evaluation of the Effect of Ultrasound-guided PENG Block on Postoperative Analgesia Management in Patients Undergoing Transcatheter Aortic Valve Implantation: A Randomized, Prospective Study
Brief Title: PENG Block forTranscatheter Aortic Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 32
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Stenosis; Aortic Diseases
Keywords: Aortic valve stenosis; Transcatheter aortic valv implantation (TAVI); PENG block; Postoperative analgesia management
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Diseases

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 20-95 years old with American Society of Anesthesiologists (ASA) classification I-IV and scheduled for TAVI will be included in the study. Patients will be randomly divided into two groups (Group PENG = PENG block group, Group Control = local infiltration group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PENG = PENG block (Active Comparator): PENG block will be performed
  Interventions: Drug: Postoperative analgesia management; Drug: PENG-Bupivacaine
- Group C = Control group (Other): Local infiltration will be applied.
  Interventions: Drug: Postoperative analgesia management; Drug: Local infiltration-Bupivacaine

INTERVENTIONS:
Drug: Postoperative analgesia management — Intravenous 0.5 mg/kg tramodol and 1 gr paracetamol will be administered to all patients 30 minutes before the end of the surgical procedure. In the postoperative period, patients will be administered iparacetamol iv 1 gr 3x1. Postoperative patient evaluation will be performed by another pain nurse who is unaware of the procedure. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic.
Drug: PENG-Bupivacaine — The probe will be placed on the anterior inferior iliac crest in the transverse plane. Then, the pubic ramus will be visualized by rotating 45 degrees. The femoral artery, iliopubic process, and psoas muscle will be visualized. The needle will be punctured with the in-plane method to reach between the pubic ramus and the psoas tendon. After the block area is confirmed with 5 ml of saline, 30 ml of local anesthetic solution containing 0.25% bupivacaine will be injected.
  Arms: Group PENG = PENG block
Drug: Local infiltration-Bupivacaine — Local infiltration will be applied with 30 ml of a local anesthetic solution containing 0.25% bupivacaine by the surgical team
  Arms: Group C = Control group

SUMMARY:
Pericapsular nerve group (PENG block) is a new fascial block defined by Arango et al. This block aims to block the femoral nerve and the accessory obturator nerve by injecting local anesthetic between the pubic ramus and psoas tendon. By blocking these nerves, anterior hip analgesia is created. It is a safe and effective method as it is applied superficially and under ultrasound guidance. In radiological and cadaver studies, it has been reported that when high volume is applied, total hip analgesia can be achieved by blocking the lateral femoral cutaneous, genitofemoral, obturator, and femoral nerves.

DETAILED DESCRIPTION:
Aortic valve stenosis (AS) is the most common valve pathology, affecting 2% to 4% of patients over the age of 75. Surgical aortic valve replacement (SAVR) has been accepted as a class I recommendation for the treatment of AS for decades. However, given that advanced age, frailty, and significant comorbidities are increasingly common in affected patients; More than one-third of high-risk and severely symptomatic AS patients are physiologically unsuitable for major surgery. This is the development and implementation of TAVI, an appropriate intervention for high-risk patients and those deemed unsuitable for surgery. With a shift in the clinical paradigm towards minimally invasive procedures, the development of TAVI has revolutionized clinical outcomes in AS, particularly in those once considered inoperable.

Selective candidate criteria and advances in operative techniques within TAVI are major contributors to successful outcomes. Basically, there are both retrograde and anterograde operative approaches that can be adopted within a TAVI procedure. While the transfemoral approach remains the most widely used, others include the transapical, transaxillary, transported, and transaortic pathways. The choice of technique adopted is greatly influenced by patient-related factors such as anatomical considerations and comorbidities present.

Because of the increasing use of ultrasound (US) in anesthesia practice, nerve blocks with US guidance are widely used. Pericapsular nerve group (PENG block) is a new fascial block defined by Arango et al. This block aims to block the femoral nerve and the accessory obturator nerve by injecting local anesthetic between the pubic ramus and psoas tendon. By blocking these nerves, anterior hip analgesia is created. It is a safe and effective method as it is applied superficially and under ultrasound guidance. In radiological and cadaver studies, it has been reported that when high volume is applied, total hip analgesia can be achieved by blocking the lateral femoral cutaneous, genitofemoral, obturator, and femoral nerves.

This prospective, randomized study, it was aimed to evaluate the efficacy of the PENG block for the management of analgesia during and after the procedure in patients undergoing TAVI. Our primary aim is to evaluate pain scores (Numerical Rating Scale-NRS), our secondary aim is to evaluate the amount of additional sedation intraoperatively, the degree of quadriceps motor block (paresis or paralysis in knee extension), and opioid-related side effects (allergic reaction, nausea, vomiting, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III,
* Aged 20-80 years
* Who will be scheduled for TAVI.

Exclusion Criteria:

* Patients who have a history of bleeding diathesis,
* Take anticoagulant therapy,
* History of chronic pain before surgery,
* Multiple trauma,
* Who cannot assess their pain (dementia),
* Who have been operated under spinal or epidural anesthesia,
* Who have an infection in the area and do not accept the procedure

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
The need for fentanyl during the procedure | Intraoperative period
  Intraoperative additional fentanyl need and dosage will be recorded

SECONDARY OUTCOMES:
Quadriceps muscle strength | Postoperative 24 hours period
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the Oxford muscle strength rating
The use of rescue analgesia | Postoperative 24 hours period]
  Meperidine using
Pain scores (Numerical Rating Scale-NRS) | Changes from baseline pain scores at postoperative 0, 2, 4, 8, 16 and 24 hours
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD

REFERENCES:
- [Background] Clayton B, Morgan-Hughes G, Roobottom C. Transcatheter aortic valve insertion (TAVI): a review. Br J Radiol. 2014 Jan;87(1033):20130595. doi: 10.1259/bjr.20130595. Epub 2013 Nov 20. PMID 24258463
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Ahiskalioglu A, Aydin ME, Ahiskalioglu EO, Tuncer K, Celik M. Pericapsular nerve group (PENG) block for surgical anesthesia of medial thigh. J Clin Anesth. 2020 Feb;59:42-43. doi: 10.1016/j.jclinane.2019.06.021. Epub 2019 Jun 15. No abstract available. PMID 31212123
- [Background] Ciftci B, Ahiskalioglu A, Altintas HM, Tekin B, Sakul BU, Alici HA. A possible mechanism of motor blockade of high volume pericapsular nerve group (PENG) block: A cadaveric study. J Clin Anesth. 2021 Nov;74:110407. doi: 10.1016/j.jclinane.2021.110407. Epub 2021 Jun 24. No abstract available. PMID 34175637
- [Derived] Gul YG, Alver S, Ozen V, Golboyu BE, Ciftci B. Pericapsular nerve group block reduces fentanyl use in transcatheter aortic valve implantation: a randomized prospective study. Clin Res Cardiol. 2025 Nov 24. doi: 10.1007/s00392-025-02815-0. Online ahead of print. PMID 41284052